CLINICAL TRIAL: NCT06239857
Title: Evaluation of the Effect of Epidural Pulsed Radiofrequency Treatment on Pain in Patients Diagnosed With Failed Back Surgery Syndrome (Persistant Spinal Pain Syndrome)
Brief Title: Epidural Pulsed Radiofrequency Treatment in Failed Back Surgery Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Principal Investigator, Burak Erken, Dr., Başakşehir Çam & Sakura City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 27.12.2023.700
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Back Pain; Failed Back Surgery Syndrome; Neuropathic Pain
MeSH Terms: conditions — Back Pain; Failed Back Surgery Syndrome; Neuralgia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidural pulsed radiofrequency treatment (Experimental): All patients diagnosed with failed back surgery syndrome will receive epidural pulsed radiofrequency treatment.
  Interventions: Procedure: Epidural pulsed radiofrequency

INTERVENTIONS:
Procedure: Epidural pulsed radiofrequency — The radiofrequency treatment is applied under sterile conditions in the operating room environment. The target epidural area is reached under fluoroscopy guidance using a radiofrequency needle. After control of the needle position, radiofrequency treatment is given. Radiofrequency parameters are set as maximum temperature 42 degrees, 45 volts, duration 6 minutes, pulse rate 2 hertz and pulse width 20 milliseconds.

SUMMARY:
Low back pain can persist in some patients with history of back surgery. In some cases, an increase in pain may even occur, and chronic pain may make treatment more difficult. A component of chronic pain is neuropathic pain, and its specific evaluation and treatment is important. Low back pain and radicular pain in the lower extremities are the main symptoms of failed back surgery syndrome (also called persistent spinal pain syndrome in new terminology).

There are many methods for treatment of failed back surgery syndrome, such as analgesic medications, physical therapy, interventional pain treatment applications, and re-surgery options. Epidural pulsed radiofrequency therapy has recently become popular among interventional pain management procedures, and studies on its effectiveness are increasing. However, studies with a multifaceted approach that also evaluate neuropathic pain are lacking in the literature. In this study, it was planned to investigate the effect of epidural pulsed radiofrequency therapy on pain palliation, including neuropathic pain, in patients diagnosed with failed back surgery syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-80
* History of at least one operation due to lumbar disc herniation
* Having radicular pain radiating to the lower extremities

Exclusion Criteria:

* Having undergone surgery for an etiology other than lumbar disc herniation
* Accompanying spinal stenosis and spondylolisthesis
* Presence of fracture, infection, coagulopathy and pregnancy
* Mental disorders that may negatively affect cooperation during assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity score | A single point in time (pre-procedural time)
  Pain severity is evaluated by using Numerical Rating Scale (NRS). In evaluation, the patient scores the pain intensity between 0 (no pain) and 10 (worst pain). It is easy to apply and takes a short time.
Change in pain severity score | A single point in time (post-procedural 1.month)
  Pain severity is evaluated by using Numerical Rating Scale (NRS). In evaluation, the patient scores the pain intensity between 0 (no pain) and 10 (worst pain). It is easy to apply and takes a short time.
Change in pain severity score | A single point in time (post-procedural 3.month)
  Pain severity is evaluated by using Numerical Rating Scale (NRS). In evaluation, the patient scores the pain intensity between 0 (no pain) and 10 (worst pain). It is easy to apply and takes a short time.
Change in pain severity score | A single point in time (post-procedural 6.month)
  Pain severity is evaluated by using Numerical Rating Scale (NRS). In evaluation, the patient scores the pain intensity between 0 (no pain) and 10 (worst pain). It is easy to apply and takes a short time.
Change in pain severity score | A single point in time (post-procedural 12.month)
  Pain severity is evaluated by using Numerical Rating Scale (NRS). In evaluation, the patient scores the pain intensity between 0 (no pain) and 10 (worst pain). It is easy to apply and takes a short time.
Change in the number of patients with neuropathic pain | A single point in time (pre-procedural time)
  The presence of neuropathic pain is assessed by Doleur Neuropathique-4 (DN-4) Questionnaire. It consists of two parts, including a physician examination part and a neuropathic pain related findings part in which the patients are questioned. A score above 4 indicates the presence of neuropathic pain.
Change in the number of patients with neuropathic pain | A single point in time (post-procedural 1.month)
  The presence of neuropathic pain is assessed by Doleur Neuropathique-4 (DN-4) Questionnaire. It consists of two parts, including a physician examination part and a neuropathic pain related findings part in which the patients are questioned. A score above 4 indicates the presence of neuropathic pain.
Change in the number of patients with neuropathic pain | A single point in time (post-procedural 3.month)
  The presence of neuropathic pain is assessed by Doleur Neuropathique-4 (DN-4) Questionnaire. It consists of two parts, including a physician examination part and a neuropathic pain related findings part in which the patients are questioned. A score above 4 indicates the presence of neuropathic pain.
Change in the number of patients with neuropathic pain | A single point in time (post-procedural 6.month)
  The presence of neuropathic pain is assessed by Doleur Neuropathique-4 (DN-4) Questionnaire. It consists of two parts, including a physician examination part and a neuropathic pain related findings part in which the patients are questioned. A score above 4 indicates the presence of neuropathic pain.
Change in the number of patients with neuropathic pain | A single point in time (post-procedural 12.month)
  The presence of neuropathic pain is assessed by Doleur Neuropathique-4 (DN-4) Questionnaire. It consists of two parts, including a physician examination part and a neuropathic pain related findings part in which the patients are questioned. A score above 4 indicates the presence of neuropathic pain.

CONTACTS AND LOCATIONS:
Overall Officials: Günay Yolcu, MD, Principal Investigator — Başakşehir Çam & Sakura City Hospital

REFERENCES:
- [Derived] Erken B, Yolcu G, Saracoglu TT. Efficacy of Epidural Pulsed Radiofrequency Treatment in Persistent Spinal Pain Syndrome: A Prospective Clinical Study. Pain Res Manag. 2025 Apr 11;2025:6200102. doi: 10.1155/prm/6200102. eCollection 2025. PMID 40255928